CLINICAL TRIAL: NCT06898723
Title: The Preventive Effect of Shenfu Injection on Myocardial Dysfunction in Sepsis: a Multicenter, Randomized Controlled Study
Brief Title: The Preventive Effect of Shenfu Injection on Myocardial Dysfunction in Sepsis
Acronym: SHIELD Trail
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: First Affiliated Hospital of Wannan Medical College (Other)
Collaborators: Suzhou Municipal Hospital of Anhui Province (Other); the Second of Affiliated Hospital of Wannan Medical College, Wuhu, China (Unknown); Wuhu County Traditional Chinese Medicine Hospital (Other); Wuhu first people's hospital (Unknown); Wuhu City Second People's Hospital (Other); Xuancheng people's hospital (Unknown); Tongling People's Hospital (Other Government); The Second Hospital of Anhui Medical University (Other); The Fourth Affiliated Hospital of Anhui Medical University (Other); The First Affiliated Hospital of Anhui Medical University (Other); The Third People's Hospital of Bengbu (Other Government); Fuyang people's hospital (Other); Chaohu Hospital of Anhui Medical University (Other); The First People's Hospital of Bengb (Unknown); Guangde people's hospital (Unknown); Fuyang Traditional Chinese Medicine Hospital (Unknown); Taihe County Traditional Chinese Medicine Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024109
Record Dates: First submitted 2025-03-15; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Septic Cardiomyopathy; Septic Shock
Keywords: Septic Shock; Cardiac Dysfunction; Shenfu Injection; Myocardial Protection; Randomized Controlled Trial
MeSH Terms: conditions — Shock, Septic | interventions — Shen-Fu

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: In this clinical trial, in addition to the ultrasound assessors mentioned above, other members of the research team, including data analysts and study coordinators, will also be masked. These individuals will not have access to specific group assignment information during the trial to ensure the objectivity of data analysis and the reliability of the results. Furthermore, participants and their immediate family members will be informed about the basic aspects of the trial but will not be disclosed the specific treatment group assignments to minimize potential bias and influence. All randomization information will be managed by an independent randomization center to ensure the integrity of the masking process.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Shenfu Injection Group (Experimental): Treatment will be conducted in accordance with international and Chinese guidelines for sepsis. On this basis, Shenfu Injection will be administered at a dosage of 50-100 ml (according to the medication practices of each participating center), diluted with an equal volume of 5% glucose and infused intravenously twice a day
  Interventions: Drug: Shenfu Injection
- Control Group (No Intervention): Treatment will be conducted in accordance with international and Chinese guidelines for sepsis.

INTERVENTIONS:
Drug: Shenfu Injection — The treatment will utilize Ginseng and Aconite Injection, which primarily consists of Red Ginseng and Aconite
  Arms: Shenfu Injection Group

SUMMARY:
This study focuses on improving heart function in patients with life-threatening blood infections (septic shock). When the body fights severe infections, the heart sometimes struggles to pump blood effectively, which can lead to dangerous complications. Current treatments like intravenous fluids and blood pressure medications have limitations in protecting heart function.

This multicenter clinical trial aims to evaluate whether adding Shenfu Injection - a traditional Chinese medicine preparation widely used to enhance cardiac function in cardiovascular diseases - to standard therapies can:

1. Prevent myocardial dysfunction during septic shock
2. Accelerate cardiac recovery if complications occur
3. Improve overall survival and clinical outcomes The randomized controlled design will compare therapeutic effects between two groups: one receiving standard septic shock treatment alone, and the other receiving standard treatment combined with Shenfu Injection.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients clinically diagnosed with septic shock must meet the diagnostic criteria of Sepsis 3.0;
* 2. Age ≥ 18 years.

Exclusion Criteria:

* 1. Pregnant or breastfeeding women;
* 2. Individuals with a history of allergies or known hypersensitivity to Ginseng and Aconite Injection or its components;
* 3. Severe underlying diseases that may affect prognosis, including uncontrolled malignant tumors with multiple metastases that are unresectable, hematological disorders, cachexia, persistent active bleeding, severe malnutrition, HIV, etc.;
* 4. Severe cardiac conditions within the last three months, including acute unstable myocardial infarction, dilated cardiomyopathy, acute coronary syndrome, acute or chronic valvular heart disease, and congestive heart failure (New York Heart Association [NYHA] Class IV);
* 5. Any of the following medical procedures performed within the last three months: any form of cardiac surgery, thoracotomy, external cardiac compression, defibrillation, direct current cardioversion, or trauma;
* 6. Use of Ginseng and Aconite Injection for less than 48 hours;
* 7. Patients expected to die within 48 hours;
* 8. Patients deemed unsuitable for this study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of septic cardiomyopathy | Day 7
Duration of vasopressor administration | 28 days
  The duration of vasopressor administration refers to the total time a patient requires vasopressor medications, measured in hours or days, to maintain blood pressure and support circulation.

SECONDARY OUTCOMES:
The incidence of septic cardiomyopathy | Day 3
Improvement in Sequential Organ Failure Assessment (SOFA) score | Day 3
  The SOFA score is used to assess and track the degree of organ dysfunction in critically ill patients. It evaluates six organ systems: respiratory, cardiovascular, hepatic, renal, coagulation, and neurological. Each organ system is scored from 0 to 4, with 0 indicating normal function and 4 indicating the most severe dysfunction. The total SOFA score ranges from 0 to 24, with higher scores indicating more severe organ dysfunction.
Improvement in Sequential Organ Failure Assessment (SOFA) Score | Day 7
  The SOFA score is used to assess and track the degree of organ dysfunction in critically ill patients. It evaluates six organ systems: respiratory, cardiovascular, hepatic, renal, coagulation, and neurological. Each organ system is scored from 0 to 4, with 0 indicating normal function and 4 indicating the most severe dysfunction. The total SOFA score ranges from 0 to 24, with higher scores indicating more severe organ dysfunction.
Fluid Balance (Total Fluid Intake and Output Measurement in Milliliters) | 3 days
  Fluid balance will be assessed by measuring total fluid intake and output in milliliters over a specified time frame. Intake includes oral and intravenous fluids, while output includes urine output, and drainage. The net fluid balance will be calculated as intake minus output, providing an indication of fluid status and potential fluid overload or deficit.
Fluid Balance (Total Fluid Intake and Output Measurement in Milliliters) | 7 days
  Fluid balance will be assessed by measuring total fluid intake and output in milliliters over a specified time frame. Intake includes oral and intravenous fluids, while output includes urine output, and drainage. The net fluid balance will be calculated as intake minus output, providing an indication of fluid status and potential fluid overload or deficit.
Duration of mechanical ventilation | 28 days
  The duration of mechanical ventilation is the total time a patient is on a ventilator, measured from initiation to extubation or removal. It reflects the severity of respiratory failure and recovery progress.
Length of Intensive Care Unit(ICU) stay | 28 days
  The length of ICU stay refers to the total duration a patient spends in the Intensive Care Unit, measured in days. It indicates the severity of the patient's condition and recovery progress.
Length of hospital stay | 28 days
  The length of hospital stay refers to the total duration a patient remains in the hospital, measured in days, from admission to discharge. It reflects the overall recovery time and treatment needs.
28-day mortality rate | 28 days
  The 28-day mortality rate refers to the percentage of patients who die within 28 days of admission, including those who are classified as deceased due to withdrawal of treatment or discharge against medical advice.
7-day mortality rate | 7 days
  The 7-day mortality rate refers to the percentage of patients who die within 7 days of admission, including those who are classified as deceased due to withdrawal of treatment or discharge against medical advice.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Wannan Medical College (Yijishan Hospital of Wannan Medical College), Wuhu, Anhui, China

IPD SHARING:
Plan to Share IPD: Yes